CLINICAL TRIAL: NCT00813670
Title: Phase 1, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of XPF-001 and to Investigate the Effect of Food on the Pharmacokinetics of a Single Dose of XPF-001 in Healthy Subjects
Brief Title: Single and Multiple Ascending Dose Safety Study of XPF-001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Dr. Paul Goldberg, Senior Director Clinical Biology and Target Discovery, Xenon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPF-001-101
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Human Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Cohort 1: Single dose of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort 2: Single dose of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort 3: Single dose of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort 4: Single dose of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort 5: Single dose of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort A: Repeated doses of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort B: Repeated doses of XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Cohort C: Repeated doses of XPF-001 (Experimental)
  Interventions: Drug: XPF-001

INTERVENTIONS:
Drug: XPF-001 — Single oral dose, or 6 days of repeated oral doses.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of single and multiple doses of XPF-001 in healthy volunteers.

The effect of food on the pharmacokinetics of XPF-001 will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (Females of non-childbearing potential) with normal or clinically insignificant laboratory results, ECGs and physical examinations.

Exclusion Criteria:

* Subjects with a presence or history of any clinically significant disease.
* Subjects who have participated in and investigational drug trial within 60 days of admission.
* Subjects who have used tobacco or nictoine products in the 1 month prior to admission
* Females who are pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
ECGs, Telemetry, Vital Signs, Physical Examinations, Laboratory Assessments and Adverse Events. | up to 14 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm, Montreal, Quebec, Canada